CLINICAL TRIAL: NCT00488046
Title: Phase I Inpatient Study of the Safety and Immunogenicity of Live Influenza A Vaccine Modified H5N1 (6-2) AA ca Recombinant (A/Hong Kong/213/2003 x A/AnnArbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for Prevention of Avian Influenza H5N1 Infection in the Event of a Pandemic
Brief Title: Single Group Study of the Safety of and Immune Response to a Bird Flu Virus Vaccine (H5N1) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 239
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Influenza; Virus Diseases
Keywords: Bird Flu
MeSH Terms: conditions — Influenza, Human; Virus Diseases; Influenza in Birds

ARMS (1):
- 1 (Experimental): Two, 0.5 ml doses of vaccine in nasal spray form administered at study entry and sometime between 4 and 8 weeks after initial vaccination
  Interventions: Biological: H5N1 (6-2) AA ca Recombinant (A/Hong Kong/213/2003 x A/AnnArbor/6/60 ca)

INTERVENTIONS:
Biological: H5N1 (6-2) AA ca Recombinant (A/Hong Kong/213/2003 x A/AnnArbor/6/60 ca) — Intranasal vaccine

SUMMARY:
Over the past decade, avian influenza (AI) has become a major health concern. The development of a safe and effective vaccine against H5N1 infection is important. The purpose of this study is to determine the safety of a new AI vaccine in healthy adults.

DETAILED DESCRIPTION:
According to the World Health Organization, the current pandemic risk associated with avian influenza H5N1 infection is serious, as an increasing number of humans are infected. Currently, H5N1 influenza transmission occurs in humans when they are exposed through direct contact to infected poultry or surfaces and objects contaminated by infected poultry feces. A pandemic occurs when a new influenza subtype emerges that infects humans, causes serious illness, and spreads easily among humans. The development of a safe and effective vaccine is necessary, should a pandemic occur. The purpose of this study is to evaluate the safety and immunogenicity of a live, attenuated A1 virus vaccine, H5N1 (6-2) AA ca Recombinant (A/Hong Kong/213/2003 x A/AnnArbor/6/60 ca).

This study will last approximately 16 weeks. Participation in this study includes a hospital stay in an isolation unit at the Johns Hopkins Bayview Medical Center. All participants will receive two doses of vaccine in nasal spray form, at study entry and sometime between 4 and 8 weeks after initial vaccination. Participants will be admitted to the isolation unit 2 days prior to each vaccination. A targeted physical exam will occur daily following each vaccination until discharge. Participants will not be discharged until nasal washes are negative. Vital signs measurement will be done at least twice daily for the duration of the inpatient stay. A follow-up outpatient visit will occur approximately 4 weeks following each vaccination. Blood and urine collection will occur at selected timepoints throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Available for the duration of the study
* Willing to use acceptable forms of contraception for the duration of the study

Exclusion Criteria:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may affect study participation
* Medical, work, or family problems as a result of alcohol or illicit drug use within 12 months prior to study entry
* Previously enrolled in an H5N1 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H5N1 influenza A virus (serum hemagglutination inhibitor [HI] titer greater than 1:8)
* Illegal drug use or dependency determined by urine test
* History of severe allergic reaction
* Allergy to oseltamivir
* Asthma or reactive airways disease within 2 years prior to study entry
* History of Guillain-Barre syndrome
* HIV infected
* Hepatitis C virus infected
* Positive for hepatitis B surface antigen (HBsAg)
* Known immunodeficiency syndrome
* Use of corticosteroid or immunosuppressive drugs within 30 days prior to vaccination. Participants who have used topical corticosteroids are not excluded.
* Live vaccines within 4 weeks prior to study vaccination
* Killed vaccines within 2 weeks prior to study vaccination
* Absence of spleen
* Blood products within 6 months prior to study vaccination
* Current smoker unwilling to stop smoking for the duration of the study
* Have traveled to the Southern Hemisphere or Asia within 14 days prior to study vaccination
* Have traveled on a cruise ship within 14 days prior to study vaccination
* Work in the poultry industry
* Other investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs or egg products
* Purified protein derivative (PPD) positive (positive tuberculosis [TB] test)
* Have family member with immunodeficiency-related condition
* Other condition that, in the opinion of the investigator, may interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Safety, defined as the frequency of vaccine-related reactogenicity events | During the acute monitoring (in-patient) phase of the study

SECONDARY OUTCOMES:
Immunogenicity, determined by anti-H5N1 antibody titer | At Days 0, 7, 9, and 28 with respect to vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cinatl J Jr, Michaelis M, Doerr HW. The threat of avian influenza A (H5N1). Part IV: Development of vaccines. Med Microbiol Immunol. 2007 Dec;196(4):213-25. doi: 10.1007/s00430-007-0052-3. Epub 2007 Jun 1. PMID 17541633
- [Background] Cox MM. Vaccines in development against avian influenza. Minerva Med. 2007 Apr;98(2):145-53. PMID 17519856
- [Background] Peiris JS, Yu WC, Leung CW, Cheung CY, Ng WF, Nicholls JM, Ng TK, Chan KH, Lai ST, Lim WL, Yuen KY, Guan Y. Re-emergence of fatal human influenza A subtype H5N1 disease. Lancet. 2004 Feb 21;363(9409):617-9. doi: 10.1016/S0140-6736(04)15595-5. PMID 14987888
- [Background] Rajagopal S, Treanor J. Pandemic (avian) influenza. Semin Respir Crit Care Med. 2007 Apr;28(2):159-70. doi: 10.1055/s-2007-976488. PMID 17458770
- [Background] Ungchusak K, Auewarakul P, Dowell SF, Kitphati R, Auwanit W, Puthavathana P, Uiprasertkul M, Boonnak K, Pittayawonganon C, Cox NJ, Zaki SR, Thawatsupha P, Chittaganpitch M, Khontong R, Simmerman JM, Chunsutthiwat S. Probable person-to-person transmission of avian influenza A (H5N1). N Engl J Med. 2005 Jan 27;352(4):333-40. doi: 10.1056/NEJMoa044021. Epub 2005 Jan 24. PMID 15668219
- [Derived] Karron RA, Talaat K, Luke C, Callahan K, Thumar B, Dilorenzo S, McAuliffe J, Schappell E, Suguitan A, Mills K, Chen G, Lamirande E, Coelingh K, Jin H, Murphy BR, Kemble G, Subbarao K. Evaluation of two live attenuated cold-adapted H5N1 influenza virus vaccines in healthy adults. Vaccine. 2009 Aug 6;27(36):4953-60. doi: 10.1016/j.vaccine.2009.05.099. Epub 2009 Jun 21. PMID 19540952